CLINICAL TRIAL: NCT04291027
Title: Comparison of Aquatic and Land-based Group Exercise for Individuals With Parkinson Disease
Brief Title: Aquatic Group Exercise for People With Parkinson Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study needed to be stopped due to the COVID-19 pandemic.
Sponsor: Ithaca College (Other)
Collaborators: Parkinson's Foundation (Other)
Responsible Party: Principal Investigator, Sarah Fishel, Assistant Professor, Ithaca College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 711
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic Group Exercise (Experimental)
  Interventions: Other: Aquatic Exercise
- Land Based Group Exercise (Active Comparator)
  Interventions: Other: Land Based Exercise

INTERVENTIONS:
Other: Land Based Exercise — Group exercise intervention will be held 2 times per week for 12 weeks and will include balance training, strengthening, gait training, and cardiovascular training.
  Arms: Land Based Group Exercise
Other: Aquatic Exercise — Group exercise intervention will be held 2 times per week for 12 weeks and will include balance training, strengthening, gait training, and cardiovascular training.
  Arms: Aquatic Group Exercise

SUMMARY:
This study will investigate the impact of land based or aquatic based group exercise on the balance, walking, balance confidence, and quality of life of people with idiopathic Parkinson disease. Participants will be randomized to participate in a land based or aquatic based group exercise program 2 times per week for 12 weeks. Prior to and after participation, balance, walking, quality of life, and balance confidence will be measured by a blinded examiner.

ELIGIBILITY:
Inclusion Criteria:

* adults over the age of 18 who have been diagnosed with idiopathic Parkinson disease.
* stable dose of levadopa medication for 30 days prior to study initiation
* able to walk 20 feet without physical assistance
* a referral from a physician to participate in physical therapy

Exclusion Criteria:

individuals with:

* uncontrolled cardiovascular or pulmonary conditions
* deep vein thrombosis in the last 6 months
* the use of breathing tube or feeding tube
* those with an extreme fear of exercising in the water
* an active dermatological condition (including eczema, psoriasis, or open wound) -any other neurological condition other than Parkinson disease
* a musculoskeletal condition that would impact their ability to participate in the exercise group
* cognitive impairment (a score of less than 24/30 on the Mini Mental Status Examination)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change in Mini-BESTest Score | Prior to intervention, after 12 week intervention
  The Mini-BESTest examines postural control. A higher scores means less balance impairment.
Change in Movement Disorder Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS): Part III | Prior to intervention, after 12 week intervention
  The Movement Disorders Society-Unified Parkinson Disease Rating Scale examines motor function for people with Parkinson disease. A higher score indicates higher motor impairment related to Parkinson disease.
Change in Gait Speed | Prior to intervention, after 12 week intervention
  The 10 meter walk test will be examined at self selected and fast speeds to examine gait speed.

SECONDARY OUTCOMES:
Change in Parkinson Disease Questionnaire-39 (PDQ-39) | Prior to intervention, after 12 week intervention
  The Parkinson disease questionnaire-39 measures quality of life for people with Parkinson disease. A higher score means more quality of life limitations related to Parkinson disease.
Change in Falls Efficacy Scale-International. | Prior to intervention, after 12 week intervention
  The Falls Efficacy Scale-International measures a person's balance confidence. A higher score is related to worse balance confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ithaca College, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886